CLINICAL TRIAL: NCT05152901
Title: A Phase 1 Comparative Bioavailability Study of Inhaled Epinephrine and Intramuscular Epinephrine Administered to Healthy Adults
Brief Title: Study of Inhaled Epinephrine and Intramuscular Epinephrine Administered to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: De Motu Cordis (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTP-00070-00
Record Dates: First submitted 2021-11-09; First posted 2021-12-10 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Anaphylactic Reaction
MeSH Terms: conditions — Anaphylaxis | interventions — Epinephrine; Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- EpiPen ®. (Active Comparator): Dosage Form- Intra muscularly (IM), Dosage- 0.3mg, Dosage Frequency and Duration- Single dose of 0.3mg epinephrine via IM on day, Visit 2.
  Interventions: Drug: EpiPen ®.
- Epinephrine (0.3mg) (Experimental): Dosage Form- Inhaled, Dosage- 0.3mg, Dosage Frequency and Duration- Single dose of 0.3mg epinephrine via inhalation on day 2 of Visit 2.
  Interventions: Drug: Epinephrine (0.3mg) inhaled
- Epinephrine (1.3mg) (Experimental): Dosage Form- Inhaled, Dosage- 1.3mg, Dosage Frequency and Duration- Single dose of 1.3mg epinephrine via inhalation on Visit 3.
  Interventions: Drug: Epinephrine (1.3mg)
- Epinephrine (4mg) (Experimental): Dosage Form- Inhaled, Dosage-4mg, Dosage Frequency and Duration- Single dose of 4mg epinephrine via inhalation on Visit 4.
  Interventions: Drug: Epinephrine (4mg)

INTERVENTIONS:
Drug: EpiPen ®. — A single dose of 0.3 mg epinephrine via intramuscular injection into the anterolateral aspect of the thigh on Day 1 Visit 2.
  Arms: EpiPen ®.
Drug: Epinephrine (0.3mg) inhaled — Participants will be administered 0.3mg of first inhaled dose of epinephrine once daily on day 2 of Visit 2
  Arms: Epinephrine (0.3mg)
Drug: Epinephrine (1.3mg) — A single inhaled dose or split into 2 administrations (administered less than 1 minute apart) of a planned dose of 1.3 mg epinephrine.
  Arms: Epinephrine (1.3mg)
Drug: Epinephrine (4mg) — A single inhaled dose or split into 2 administrations (administered less than 1 minute apart) of a planned dose of 4 mg epinephrine
  Arms: Epinephrine (4mg)

SUMMARY:
This is a study to determine the relative bioavailability of inhaled epinephrine compared with 0.3mg epinephrine administered IM in healthy male and female participants.

DETAILED DESCRIPTION:
DMC-IH1 (Investigational Product) is a capsule containing epinephrine bitartrate dry powder blend contained within a single-use, proprietary inhalation device.

The planned dosages for inhalation are 0.3 mg on Visit 2, 1.3 mg (dose will not exceed 6 mg) on Visit 3, and 4 mg (dose will not exceed 6 mg) on Visit 4.

The study will comprise 3 periods: Screening, Treatment, and Follow-up. Total duration of the study is approximately 66 days including -28 days from screening to visit to follow up

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and ≥ 18 to ≤ 45 years of age at time of signing the Informed Consent Form.
2. BMI is between ≥18.00 to 29.00 kg/m2 with a minimum body weight of 45.0 kg.
3. Participant who is in good health based on the results of medical history, physical examination, vital sign measurements, and clinical laboratory evaluations, as assessed by the Investigator (or designee) with a resting heart rate of ≤ 90 beats per minute and systolic blood pressure of ≤ 130/90 mmHg and diastolic blood pressure of ≤ 90/50 mmHg.
4. Has normal lung function assessed using spirometry and defined by FVC ≥ lower limit of normal (LLN), FEV1/FVC ≥ LLN, and PIF ≥ LLN. (FVC- Functional Vital Capacity; FEV- Forced Expiratory Volume)
5. Has no history of anaphylaxis or severe allergy requiring the use of epinephrine.
6. Who is a non-smoker; or social smoker who only used nicotine on ≤ 5 occasions within 30 days prior to Screening, a negative cotinine test at Screening, and ability and willingness to refrain from tobacco products for the duration of the study (from 7 days prior to the first dose through to EOS [Visit 5]).

Exclusion Criteria:

1. Participant who is pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study (through Visit 5/EOS).
2. Participant has a history of significant hypersensitivity or intolerance to lactose.
3. Participant has a history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee) except for fully resolved childhood asthma.
4. Participant has a positive urine drug screen (including cotinine) at Screening and at Baseline (Visit 2/Day -1).
5. Participant has a positive COVID-19 test at Screening and prior to Baseline (Visit 2/Day -1)
6. Participant took part a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives prior to Baseline (Visit 2/Day -1).
7. Participant used or intends to use any prescription or non-prescription medications/products within 14 days prior to dosing through to Follow-up (Visit 5), with the exception of Oral contraceptive pill (OCPs) and paracetamol/acetaminophen (1 therapeutic dose [1g] three times per week) at the discretion of the Investigator, and contraceptives.
8. Participant has a history of alcoholism, substance or drug abuse-related disorders deemed significant by the Investigator (or designee) (ie, > 14 drinks/week for women or > 21 drinks/week for men [1 drink = 150 mL of wine or 360 mL of beer or 45 mL of hard liquor]) within the last 3 months prior to dosing, must not have consumed more than 14 drinks per week in any week or have a history of alcohol abuse within the last 12 months.
9. Participant has a positive alcohol breath test at Screening and prior to dosing with Investigational Product (IP) at Visit 2, Visit 3, and Visit 4.
10. Female participant has a positive urine pregnancy test prior to dosing with IP at Visit 2, Visit, 3, and Visit 4.
11. Participant has a positive test for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV) with HCV RNA detected at Screening or Day 1 and hepatitis B core antibody (HBcAb) at Screening only.
12. Participant has presence of any physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the protocol or complete the study per protocol.
13. Participant has received any of the following vaccinations:

    1. Live vaccine(s) within 1 month prior to Screening or plans to receive such vaccines during the study.
    2. Killed vaccine 1 week prior to Screening.
    3. COVID-19 vaccine Day -7 through to Visit 4.
14. Participant had surgery of the nose/paranasal sinuses/mouth/throat within 8 weeks prior to Screening.
15. Participant has any clinically relevant respiratory (especially with reduction of respiratory capacity) or cardiovascular abnormality (eg, high blood pressure, myocardial infarction in previous 3 months, etc), or any other abnormality that in the opinion of the Investigator may pose a safety risk to a participant in this study, may confound the clinical performance or safety assessment, or may interfere with study participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Regulatory Activities (MedDRA) Version 22.0 or higher. | Screening through to follow up so approx. 66 days
Safety and tolerability of inhaled epinephrine in healthy participants measured through percentage of subjects with abnormal and clinically significant abnormal hematology values. | Screening through to follow up so approx. 66 days
Safety and tolerability of inhaled epinephrine in healthy participants measured through PR interval in ECG Assessment. | Screening through to follow up so approx. 66 days
  PR interval is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex (the onset of ventricular depolarization)
Change in Baseline of heart rate will be monitored from 15 minutes prior to each dosing (to establish baseline) through safety continuous cardiac monitoring (Telemetry) at timepoints to match the pharmacokinetic blood draws. | Screening through to follow up so approx. 66 days
Safety and tolerability of inhaled epinephrine in healthy participants measured through Functional Vital Capacity (FVC) in the Lung Function test assessment. | Screening through to follow up so approx. 66 days

SECONDARY OUTCOMES:
To determine the plasma pharmacokinetics (PK) of inhaled epinephrine in healthy participants through time to maximum observed epinephrine concentration (Tmax). | Day 1, Day 2, Day16 and Day 30
To determine the plasma pharmacokinetics (PK) of inhaled epinephrine in healthy participants by plasma concentration-time profiles (Cmax). | Day 1, Day 2, Day16 and Day 30
To determine the plasma pharmacokinetics (PK) of inhaled epinephrine in healthy participants through Area under curve (AUC0-t). | Day 1, Day 2, Day16 and Day 30
  Area under the drug concentration-time curve, from time zero (time of dosing) to the last time point (AUC0-t)
To determine the comparative plasma bioavailability of inhaled epinephrine to intramuscular (IM)epinephrine in healthy participants. | Day 1, Day 2, Day16 and Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Neill, Study Director — peter.oneill@demotucordis.co
Locations (1):
- Q-Pharm Pty Ltd, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No